CLINICAL TRIAL: NCT03573037
Title: Duration of Anticoagulation Therapy Following Catheter Ablation of Atrial Fibrillation; Randomized Controlled Trial
Brief Title: Anticoagulation After RFCA
Acronym: Reducible
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yong Seog Oh (Other)
Responsible Party: Sponsor-Investigator, Yong Seog Oh, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REDUCIBLE
Record Dates: First submitted 2017-04-24; First posted 2018-06-29 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Anticoagulants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1-month anticoagulation group (Experimental): Anticoagulation using warfarin or non-VKA oral anticoagulant for 1 month after radiofrequency catheter ablation of paroxismal atrial fibrillation and then stop anticoagulation.
  Interventions: Drug: Oral anticoagulant
- 2-month anticoagulation group (Active Comparator): Anticoagulation using warfarin or non-VKA oral anticoagulant for 2 months after radiofrequency catheter ablation of paroxismal atrial fibrillation and then stop anticoagulation
  Interventions: Drug: Oral anticoagulant

INTERVENTIONS:
Drug: Oral anticoagulant — 1:1 randomization to 1-month anticoagulation or 2-month anticoagulation after radiofrequency catheter ablation of paroxismal atrial fibrillation

SUMMARY:
The anticoagulation therapy is needed when rhythm control strategy is applied in atrial fibrillation patients but adverse events such as major bleeding exist. This study aims to examine the prognostic inpact of the duration of anticoagulation after radiofrequency ablation of paroxismal atrial fibrillation in patients with low thromboembolic risk. Paroxismal atrial fibrillation patients with 0 or 1 CHADS2-Vasc score undergoing radiofrequency ablation is randomized into one month anticoagulation group and two months anticoagulation group after the procedure. Thromboembolic event and adverse event including major or minor bleeding would be compared.

DETAILED DESCRIPTION:
Catheter based radiofrequency ablation has been used in more than a decade as a rhythm control therapy. Recently, superior outcome to medical therapy has been constantly reported and the radiofrequency catheter ablation (RFCA) became popular globally. It is recommended to anticoagulate patients who received RFCA for atrial fibrillation at least two months after the procedure. However, a few reports suggest anticoagulation in selective patients according to CHADS2-Vasc score. Anticoagulants prevent thromboembolic event in atrial fibrillation but the risk of bleeding is increased in company. There is controversy in the duration of anticoagulation after RFCA of atrial fibrillation. The investigators aimed to investigate the association with thromboembolic and bleeding event of anticoagulation duration after RFCA of atrial fibrillation in patients with low thromboembolic risk. Paroxismal atrial fibrillation patients with 0 or 1 CHADS2-Vasc score who are undergoing RFCA are included and randomized by 1:1 ratio to one month anticoagulation group and two months anticoagulation group after RFCA. Any patient with an evidence of intracardiac thrombus is excluded. The primary endpoint is thromboembolic event in 6 months after RFCA and the secondary endpoint is bleeding event in 6 months after RFCA.

ELIGIBILITY:
Inclusion Criteria:

* Under 75 years old Patients undergoing RFCA for paroxismal atrial fibrillation CHADS-Vasc score 0-1

Exclusion Criteria:

* Presence of intracardiac thrombus

Max Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2014-07; Primary Completion 2020-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Thromboembolic event | 6 months
  Composite of ischemic stroke, transient ischemic attack, or other systemic embolic events

SECONDARY OUTCOMES:
Major bleeding | 6 months
  bleeding events that result in a reduction in hemoglobin level of at least 20 g per liter, transfusion of at least 2 units of blood, or symptomatic bleeding in a critical area or organ

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Seog Oh, MD,PhD, Principal Investigator — The Catholic University of Korea
Locations (1):
- Seoul St Mary's Hospital, Seoul, Seo Ch-gu, South Korea